CLINICAL TRIAL: NCT00423189
Title: Lucentis Utilizing Visudyne (LUV Trial)-- Reduced Fluence Photodynamic Therapy With Visudyne Combined With Intravitreal Ranibizumab in the Treatment of Age-Related Macular Degeneration
Brief Title: Lucentis Utilizing Visudyne (LUV Trial) Combination Therapy in the Treatment of Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: David M. Brown, M.D. (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, David M. Brown, M.D., Director of Research, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUV
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Age-Related Macular Degeneration
Keywords: LUV; Lucentis; Visudyne; PDT; AMD; ARMD; Age; Related; Macular; Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; 1-phenyl-3,3-dimethyltriazene; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ranibizumab only (Active Comparator): drug - intravitreal ranibizumab
  Interventions: Drug: Ranibizumab (Lucentis); Drug: 0.5mg ranibizumab
- 40% fluence PDT/procedure (Experimental): 40% fluence photodynamic therapy-PDT therapy with 0.5mg ranibizumab
  Interventions: Drug: Ranibizumab (Lucentis); Drug: 0.5mg ranibizumab
- 20% fluence photodynamic therapy (Experimental): 20% fluence photodynamic therapy-PDT therapy with 0.5mg ranibizumab
  Interventions: Drug: Ranibizumab (Lucentis); Drug: 0.5mg ranibizumab

INTERVENTIONS:
Drug: Ranibizumab (Lucentis) — as needed, one intravitreal injection of 0.50mg ranibizumab
  Other Names: PDT; Photodynamic Therapy
Drug: 0.5mg ranibizumab — as needed, one intravitreal injection of 0.50mg ranibizumab
  Other Names: lucentis

SUMMARY:
The PDT/Lucentis trial will be a Phase IV comparative trial comparing the use of combination therapy with ITV ranibizumab and verteporfin PDT to ITV ranibizumab alone in patients with exudative AMD.

DETAILED DESCRIPTION:
The PDT/Lucentis trial will be a Phase IV comparative trial comparing the use of combination therapy with ITV ranibizumab and verteporfin PDT to ITV ranibizumab alone in patients with exudative AMD. Patients will be randomized to one of three groups. All patients will receive three consecutive monthly treatments with ITV ranibizumab. Patients randomized to group I will receive only ITV ranibizumab. Patients randomized to group II will also receive one treatment with reduced fluence (20% fluence) verteporfin PDT at day 0. Patients randomized to group III will also receive one treatment with reduced fluence (40% fluence) vPDT. All patients will also be evaluated for possible retreatment with ranibizumab according to established criteria. Thirty patients (ten per group) will be recruited from one U.S. sites in a 6-month period. Randomization will occur at the time of entry into the study. Follow-up will continue until month 12 (from day 0) in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 55 years
* Subfoveal neovascular membrane confirmed by fluorescein angiography and or ICG
* Visual acuity not better than 20/32 and not worse than 20/320 by ETDRS refraction

Exclusion Criteria:

* Any previous vitrectomy in study eye (posterior or anterior associated with vitreous loss in cataract surgery)
* Intracapsular cataract extraction (posterior capsule needs to be present)
* Previous treatment with ranibizumab
* Previous treatment with pegaptanib
* Previous treatment with ITV triamcinolone
* Any previous treatment with photodynamic therapy
* Previous history of retinal detachment in study eye
* Any previous radiation treatments to head/ neck
* Significant cardiovascular disease or cancer that would prevent follow-up visits or completion of the 12 month study
* Prior enrollment in any study for AMD in the study eye
* Participation in another simultaneous medical investigator or trial
* Ocular disorders in the study eye that may confound interpretation of study results, including retinal detachment or macular hole.
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the study period
* Aphakia or absence of the posterior capsule in the study eye
* Previous violation of the posterior capsule is also excluded unless it occurred as a result of YAG laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
* History of idiopathic or autoimmune uveitis in either eye
* Significant structural damage to the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s)
* Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by OCT
* Ocular inflammation (including trace or above) in the study eye
* Uncontrolled glaucoma (defined as intraocular pressure ≥30 mm Hg despite treatment with anti- medications) or previous filtration surgery in the study eye
* Infectious blepharitis, keratitis, scleritis, or conjunctivitis (in either eye) or current treatment for serious systemic infection
* Spherical equivalent of the refractive error in the study eye of more than -8 diopters myopia (For patients who have had refractive or cataract surgery in the study eye, pre-operative spherical equivalent refractive error of more than -8 diopters myopia is not allowed)

Systemic Conditions

* Uncontrolled Blood pressure exceeding diastolic pressure of 100 mm Hg (sitting) during the screening period
* Uncontrolled diabetes mellitus
* Renal failure requiring dialysis or renal transplant
* Premenopausal women not using adequate contraception
* Previous participation in other studies of investigational drugs (excluding vitamins and minerals) within 3 months preceding Day 0
* History of other disease, metabolic dysfunction, physical examination finding, or other findings giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications
* INR ≥ 3.0 (e.g. due to current treatment with warfarin). The use of aspirin is not an exclusion.

Other

* History of allergy to fluorescein, not amenable to treatment
* History of allergy to shellfish
* History of allergy to intravenous iodine
* History of allergy to indocyanine green
* Inability to obtain fundus photographs or angiograms of sufficient quality to be analyzed and graded by the central reading center
* Inability to comply with study or follow up procedures
* History of allergy to humanized antibodies or any component of the ranibizumab formulation

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Brown, M.D., Principal Investigator — Vitreoretinal Consultants
Locations (1):
- Vitreoretinal Consultants, Houston, Texas, United States

REFERENCES:
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Michels S, Hansmann F, Geitzenauer W, Schmidt-Erfurth U. Influence of treatment parameters on selectivity of verteporfin therapy. Invest Ophthalmol Vis Sci. 2006 Jan;47(1):371-6. doi: 10.1167/iovs.05-0354. PMID 16384987
- [Background] Azab M, Boyer DS, Bressler NM, Bressler SB, Cihelkova I, Hao Y, Immonen I, Lim JI, Menchini U, Naor J, Potter MJ, Reaves A, Rosenfeld PJ, Slakter JS, Soucek P, Strong HA, Wenkstern A, Su XY, Yang YC; Visudyne in Minimally Classic Choroidal Neovascularization Study Group. Verteporfin therapy of subfoveal minimally classic choroidal neovascularization in age-related macular degeneration: 2-year results of a randomized clinical trial. Arch Ophthalmol. 2005 Apr;123(4):448-57. doi: 10.1001/archopht.123.4.448. PMID 15824216
- See also: GreaterHRR website — http://www.houstonretina.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 patients, over a 12 month period were followed after receiving treatment of either decreased fluence(2 different fluences) and 0.5mg ranibizumab, as compared to monotherapy of 0.5mg ranibizumab at a single site
Pre-assignment Details: patients that were considered to have recalcitrant wet age related macular degeneration were recruited for this trial
Groups:
- Ranibizumab and 40% Fluence PDT(Procedure): 40% fluence photodynamic therapy - procedure
- Ranibizumab and 20% Fluence PDT(Procedure): 20% fluence photodynamic therapy - procedure
Period: Overall Study
Arm/Group | Ranibizumab Only | Ranibizumab and 40% Fluence PDT(Procedure) | Ranibizumab and 20% Fluence PDT(Procedure)
Started | 2 | 3 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: drug - intravitreal ranibizumab
- Arm 2: 40% fluence photodynamic therapy - procedure
- Arm 3: 20% fluence photodynamic therapy - procedure
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 2 | 3 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (3) | 78 (7) | 67 (5) | 72 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 3 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 2 | 03 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Best-corrected ETDRS Visual Acuity at 6 Months and 12 Months Only Time Points (Gain or Loss of >15 Letters at 12 Months)
Description: Visual Acuity was measured by ETDRS by certified refractionists in certified lanes at 12 months. Visual Acuity was not measured by ETDRS at 6 months.
Time Frame: 1 Year
Population: As per subjects participated
Measure: Number; unit: participants
Groups:
- Ranibizumab Only: IVT Ranibizumab only
- 40% Fluence PDT/Ranibizumab: 40% Fluence PDT WITH ivt Ranibizumab
- 20% Fluence PDT/Ranibizumab: 20% Fluence PDT with IVT Ranibizumab
Arm/Group | Ranibizumab Only | 40% Fluence PDT/Ranibizumab | 20% Fluence PDT/Ranibizumab
Number analyzed (Participants) | 2 | 3 | 2
participants | 0 | 0 | 0

2. Secondary Outcome: Number of Intravitreal Injections With Ranibizumab Needed by Patients at 12 Months
Description: Number of intravitreal injections with ranibizumab needed by patients at 12 months was not determined due to lack of efficacy.
Time Frame: 1 Year
Population: not determined due to lack of efficacy
Groups:
- 40% Fluence Photodynamic Therapy Combined With Ranibizumab: 40% fluence photodynamic therapy combined with ranibizumab- procedure
- 20% Fluence Photodynamic Therapy Combined With Ranibizumab: 20% fluence photodynamic therapy combined with ranibizumab- procedure
Arm/Group | Ranibizumab Only | 40% Fluence Photodynamic Therapy Combined With Ranibizumab | 20% Fluence Photodynamic Therapy Combined With Ranibizumab
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: OCT 3 Macular Thickness Improvement (Baseline-1month, 2months, 3months, 6months &12 Months)
Description: OCT 3 macular thickness improvement at Baseline-1month, 2months, 3months, 6months &12 months was not determined due to lack of efficacy.
Time Frame: 1 Year
Arm/Group | Ranibizumab Only | 40% Fluence Photodynamic Therapy Combined With Ranibizumab | 20% Fluence Photodynamic Therapy Combined With Ranibizumab
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Choroidal Perfusion as Assessed by ICG Angiography at 1, 2, 3, 6, and 12 Months
Description: Choroidal perfusion as assessed by ICG angiography at 1, 2, 3, 6, and 12 months was not determined due to lack of efficacy
Time Frame: 1 Year
Arm/Group | Ranibizumab Only | 40% Fluence Photodynamic Therapy Combined With Ranibizumab | 20% Fluence Photodynamic Therapy Combined With Ranibizumab
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Safety of Combination Therapy With Verteporfin PDT and ITV Ranibizumab
Description: Safety of combination therapy with verteporfin PDT and ITV ranibizumab was not determined due to lack of efficacy.
Time Frame: 1 Year
Groups:
- 40% Fluence Photodynamic Therapy Combined With Ranibizumab: 40% fluence photodynamic therapy/combined with ranibizumab - procedure
- 20% Fluence Photodynamic Therapy Combined With Ranibizumab: 20% fluence photodynamic therapy combined with ranibizumab - procedure
Arm/Group | Ranibizumab Only | 40% Fluence Photodynamic Therapy Combined With Ranibizumab | 20% Fluence Photodynamic Therapy Combined With Ranibizumab
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Ranibizumab Only: subject only received ranibizumab
- 40% Fluence PDT Combined With Ranibizumab: Subjects who have received 40% fluence PDT combined with as needed dosing with ranibizumab
- 20% PDT Fluence Combined With Ranibizumab: Subjects who received 20% with as needed ranibizumab
Arm/Group | Ranibizumab Only | 40% Fluence PDT Combined With Ranibizumab | 20% PDT Fluence Combined With Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/3 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab Only (N=2) | 40% Fluence PDT Combined With Ranibizumab (N=3) | 20% PDT Fluence Combined With Ranibizumab (N=2)
Death of unknown origin (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab Only (N=2) | 40% Fluence PDT Combined With Ranibizumab (N=3) | 20% PDT Fluence Combined With Ranibizumab (N=2)
1+ Nuclear Sclerosis (Eye disorders) | 1 (2) | 1 (3) | 1 (2) — The cataract changes were found on a slip lamp/anterior chamber evaluation.
2+ nuclear sclerosis (Eye disorders) | 1 (2) | 1 (3) | 1 (2)

LIMITATIONS AND CAVEATS:
The trial was discontinued due to a lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes